CLINICAL TRIAL: NCT03815656
Title: An Integrated Biomarker Approach to Personalized, Adaptive Deep Brain Stimulation in Parkinson Disease [Formerly: Scalar Closed-Loop STN/GPi DBS Based on Evoked and Spontaneous Potentials (Permanently Implanted Medtronic RC+S Studies)]
Brief Title: Closed Loop DBS Implanted RC+S Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dennis Turner, M.D. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Duke University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Dennis Turner, M.D., Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100982; UH3NS103468 (NIH); UH3NS129898 (NIH)
Record Dates: First submitted 2019-01-17; First posted 2019-01-24 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Implanted RC+S (Experimental): Implanted Medtronic RC+S IPG with dual DBS electrodes in STN and GPi. DBS stimulation will be administered to: 1) STN alone, 2) GPi alone, 3) cooperative STN + GPi, and 4) adaptive, closed-loop stimulation of STN and/or GPi.
  Interventions: Device: STN alone; Device: GPi alone; Device: STN + GPi; Device: Closed-loop stimulation

INTERVENTIONS:
Device: STN alone — DBS stimulation of STN alone
Device: GPi alone — DBS stimulation of GPi alone
Device: STN + GPi — cooperative DBS stimulation of STN and GPi sites
Device: Closed-loop stimulation — adaptive DBS stimulation of STN and/or GPi sites

SUMMARY:
This study involves patients who are already planning to have deep brain stimulation (DBS) surgery to treat the symptoms of severe Parkinson's Disease (PD). The study has two goals:

1. to evaluate the effectiveness of implanting DBS electrodes in the two most common locations for DBS (subthalamic nucleus (STN), and globus pallidus interna (GPi)), instead of just one electrode, on each side of the brain; and
2. to develop an adaptive DBS system using brain signals measured from these two electrodes.

DETAILED DESCRIPTION:
The purpose of this study is a small, first in man, clinical feasibility trial for patients with severe Parkinson's Disease (PD), who are already clinically eligible for deep brain stimulation (DBS) with two goals:

1. to compare efficacy from two common sites of DBS (subthalamic nucleus (STN), and globus pallidus interna (GPi)) through the implantation of dual DBS electrodes on each side of the brain; and
2. to develop a closed loop DBS system using evoked and spontaneous potentials derived from these two electrodes.

The study will involve bilateral dual DBS electrode placement in clinically standard locations (ie, STN and GPi) unilaterally or (more often) bilaterally, the placement of the RC+S Medtronic research implantable pulse generator (IPG), and a commitment to return for both extensive postoperative programming and testing to define clinical efficacy and separate research days to develop the closed loop approach. In addition, patients will undergo intraoperative research using temporary percutaneous extensions to the DBS electrode(s) and DBS lead cannula after implantation to confirm the electrode location and to identify what the signals will look like during later chronic recordings through the research IPG.

The research RC+S IPG includes both ordinary DBS stimulation as well as a recording system that simultaneously measures the DBS local evoked potential (DLEP) and/or local field potential (LFP) responses from either the same or a second DBS electrode.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* diagnosed with Parkinson's Disease and is considered a surgical candidate for DBS
* has medication-related side effects from levodopa (i.e., dyskinesias, on-off fluctuations)
* has off-on improvement with levodopa of at least 30%
* is available for follow-up visits for length of study

Exclusion Criteria:

* is not safe surgical candidate for DBS
* has severe neurological injury or disease other than Parkinson's Disease
* has condition requiring repeated MRI scans
* has untreated, clinically significant depression
* has an electrical or electromagnetic implant
* had a prior thalamotomy or surgical ablation procedure
* has dementia interfering with ability to comply with study requirements or give informed consent
* abuses drugs or alcohol
* has a history of seizures
* has any metallic implants
* is pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) score: "on" medication, "on" stimulation at 12 months after IPG implant. | baseline and 12 months after IPG implant
  Change in UPDRS score for subject from baseline (pre-surgery) "on" medication state to "on" medication and "on" stimulation state at 12 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. The scores from four subscales (1. Mentation, Behavior and Mood, 2. Activities of Daily Living, 3. Motor Examination, and 4. Complications of Therapy) are summed to determine the total UPDRS score. Total scores range from 0 (no disability) to 199 (total disability).
Change in Unified Parkinson's Disease Rating Scale (UPDRS) score: "on" medication, "on" stimulation at 24 months after IPG implant. | baseline and 24 months after IPG implant
  Change in UPDRS score for subject from baseline (pre-surgery) "on" medication state to "on" medication and "on" stimulation state at 24 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. The scores from four subscales (1. Mentation, Behavior and Mood, 2. Activities of Daily Living, 3. Motor Examination, and 4. Complications of Therapy) are summed to determine the total UPDRS score. Total scores range from 0 (no disability) to 199 (total disability).
Change in Unified Parkinson's Disease Rating Scale (UPDRS) score: "on" medication, "on" stimulation at 48 months after IPG implant. | baseline and 48 months after IPG implant
  Change in UPDRS score for subject from baseline (pre-surgery) "on" medication state to "on" medication and "on" stimulation state at 48 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. The scores from four subscales (1. Mentation, Behavior and Mood, 2. Activities of Daily Living, 3. Motor Examination, and 4. Complications of Therapy) are summed to determine the total UPDRS score. Total scores range from 0 (no disability) to 199 (total disability).
Change in Unified Parkinson's Disease Rating Scale (UPDRS) score: "on" medication, "on" stimulation at 72 months after IPG implant. | baseline and 72 months after IPG implant
  Change in UPDRS score for subject from baseline (pre-surgery) "on" medication state to "on" medication and "on" stimulation state at 72 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. The scores from four subscales (1. Mentation, Behavior and Mood, 2. Activities of Daily Living, 3. Motor Examination, and 4. Complications of Therapy) are summed to determine the total UPDRS score. Total scores range from 0 (no disability) to 199 (total disability).

SECONDARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale, subscale III: Motor Evaluation (UPDRS-III) score: "off" medication, "on" stimulation at 12 months after IPG implant. | baseline and 12 months after IPG implant
  Change in UPDRS-III (Motor Evaluation) score from baseline (pre-surgery) "off" medication state to "off" medication and "on" stimulation state at 12 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. Subscale III, Motor Examination, scores range from 0 (no disability) to 108 (total disability).
Change in Unified Parkinson's Disease Rating Scale, subscale III: Motor Evaluation (UPDRS-III) score: "off" medication, "on" stimulation at 24 months after IPG implant. | baseline and 24 months after IPG implant
  Change in UPDRS-III (Motor Evaluation) score from baseline (pre-surgery) "off" medication state to "off" medication and "on" stimulation state at 24 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. Subscale III, Motor Examination, scores range from 0 (no disability) to 108 (total disability).
Change in Unified Parkinson's Disease Rating Scale, subscale III: Motor Evaluation (UPDRS-III) score: "off" medication, "on" stimulation at 48 months after IPG implant. | baseline and 48 months after IPG implant
  Change in UPDRS-III (Motor Evaluation) score from baseline (pre-surgery) "off" medication state to "off" medication and "on" stimulation state at 48 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. Subscale III, Motor Examination, scores range from 0 (no disability) to 108 (total disability).
Change in Unified Parkinson's Disease Rating Scale, subscale III: Motor Evaluation (UPDRS-III) score: "off" medication, "on" stimulation at 72 months after IPG implant. | baseline and 72 months after IPG implant
  Change in UPDRS-III (Motor Evaluation) score from baseline (pre-surgery) "off" medication state to "off" medication and "on" stimulation state at 72 months after IPG implant. The UPDRS is a scale to measure the degree of a patient's disability due to Parkinson's Disease. Subscale III, Motor Examination, scores range from 0 (no disability) to 108 (total disability).
Change in percentage of waking hours with good "on" time at 12 months after IPG implant. | baseline and 12 months after IPG implant
  Change in percentage of waking hours subject experienced "on" time without troubling dyskinesias, based on 3-day motor diary, compared to pre-surgery baseline.
Change in percentage of waking hours with good "on" time at 24 months after IPG implant. | baseline and 24 months after IPG implant
  Change in percentage of waking hours subject experienced "on" time without troubling dyskinesias, based on 3-day motor diary, compared to pre-surgery baseline.
Change in percentage of waking hours with good "on" time at 48 months after IPG implant. | baseline and 48 months after IPG implant
  Change in percentage of waking hours subject experienced "on" time without troubling dyskinesias, based on 3-day motor diary, compared to pre-surgery baseline.
Change in percentage of waking hours with good "on" time at 72 months after IPG implant. | baseline and 72 months after IPG implant
  Change in percentage of waking hours subject experienced "on" time without troubling dyskinesias, based on 3-day motor diary, compared to pre-surgery baseline.
Change in Parkinson's Disease Questionnaire-39 (PDQ-39) patient satisfaction score at 12 months after IPG implant. | baseline and 12 months after IPG implant
  Change in PDQ-39 score compared to pre-surgery baseline. The PDQ-39 is a 39-item self-reporting questionnaire to assess the impact of Parkinson's Disease on quality of life. The PDQ-39 is divided into 8 dimensions (1. Mobility, 2. Activities of Daily Life, 3. Emotional Well-being, 4. Stigma, 5. Social Support, 6. Cognition, 7. Communication, and 8. Bodily Discomfort). The total score is the sum of the dimension total scores divided by 8. Scores range from 0 (better quality of life) to 100 (worse quality of life).
Change in Parkinson's Disease Questionnaire-39 (PDQ-39) patient satisfaction score at 24 months after IPG implant. | baseline and 24 months after IPG implant
  Change in PDQ-39 score compared to pre-surgery baseline. The PDQ-39 is a 39-item self-reporting questionnaire to assess the impact of Parkinson's Disease on quality of life. The PDQ-39 is divided into 8 dimensions (1. Mobility, 2. Activities of Daily Life, 3. Emotional Well-being, 4. Stigma, 5. Social Support, 6. Cognition, 7. Communication, and 8. Bodily Discomfort). The total score is the sum of the dimension total scores divided by 8. Scores range from 0 (better quality of life) to 100 (worse quality of life).
Change in Parkinson's Disease Questionnaire-39 (PDQ-39) patient satisfaction score at 48 months after IPG implant. | baseline and 48 months after IPG implant
  Change in PDQ-39 score compared to pre-surgery baseline. The PDQ-39 is a 39-item self-reporting questionnaire to assess the impact of Parkinson's Disease on quality of life. The PDQ-39 is divided into 8 dimensions (1. Mobility, 2. Activities of Daily Life, 3. Emotional Well-being, 4. Stigma, 5. Social Support, 6. Cognition, 7. Communication, and 8. Bodily Discomfort). The total score is the sum of the dimension total scores divided by 8. Scores range from 0 (better quality of life) to 100 (worse quality of life).
Change in Parkinson's Disease Questionnaire-39 (PDQ-39) patient satisfaction score at 72 months after IPG implant. | baseline and 72 months after IPG implant
  Change in PDQ-39 score compared to pre-surgery baseline. The PDQ-39 is a 39-item self-reporting questionnaire to assess the impact of Parkinson's Disease on quality of life. The PDQ-39 is divided into 8 dimensions (1. Mobility, 2. Activities of Daily Life, 3. Emotional Well-being, 4. Stigma, 5. Social Support, 6. Cognition, 7. Communication, and 8. Bodily Discomfort). The total score is the sum of the dimension total scores divided by 8. Scores range from 0 (better quality of life) to 100 (worse quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Turner, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared: IPD for all participants that support the primary and secondary outcome measures listed in clinicaltrials.gov, after deidentification.
Supporting Information: ICF
Time Frame: Data are available now through the end of funding (estimated January 2027). Additional data are updated on an annual basis.
Access Criteria: Supporting Information (informed consent form) is available on clinicaltrials.gov.
  IPD are available by request at the Data Archive for the BRAIN Initiative (dabi.loni.usc.edu). Requests for access will be evaluated through the end of grant funding (estimated January 2027).
URL: https://dabi.loni.usc.edu

REFERENCES:
- [Derived] Mitchell KT, Schmidt SL, Cooney JW, Grill WM, Peters J, Rahimpour S, Lee HJ, Jung SH, Mantri S, Scott B, Lad SP, Turner DA. Initial Clinical Outcome With Bilateral, Dual-Target Deep Brain Stimulation Trial in Parkinson Disease Using Summit RC + S. Neurosurgery. 2022 Jul 1;91(1):132-138. doi: 10.1227/neu.0000000000001957. Epub 2022 Apr 7. PMID 35383660

DOCUMENTS (1):
  • Informed Consent Form (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT03815656/ICF_000.pdf